CLINICAL TRIAL: NCT00575510
Title: Intervention to Improve Follow-up of Abnormal Pap Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 05-245; R01CA107015 (NIH)
Record Dates: First submitted 2007-12-14; First posted 2007-12-18 (Estimated); Results first posted 2014-08-15 (Estimated); Last update posted 2018-08-23 (Actual); Status verified 2018-07

CONDITIONS: Cervical Cancer
Keywords: unified theory of behavior; Pap test; cervical dysplasia; women's health
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Cervical Dysplasia | interventions — Methods

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Intervention (Experimental): Culturally targeted behavioral and normative beliefs + knowledge/skills + salience + environmental constraints/barriers counseling
  Interventions: Behavioral: Intervention
- Active Control (Active Comparator): nontargeted behavioral and normative beliefs + knowledge/skills + salience + environmental constraints/barriers counseling
  Interventions: Behavioral: Active control
- Standard Care Only (No Intervention): Clinical standard of care at time of study

INTERVENTIONS:
Behavioral: Intervention — Multiple component intervention based in the unified theory of behavior
  Arms: Intervention
Behavioral: Active control — Partial intervention (full intervention minus cultural-specific component)
  Arms: Active Control

SUMMARY:
This project will examine whether a theory-based telephone intervention delivered by a nurse at the time women are informed of an abnormal Pap test result will increase adherence to follow-up recommendations.

DETAILED DESCRIPTION:
Over 90% of deaths due to cervical cancer could be prevented with appropriate screening and treatment of precursor lesions. However, 20% to 70% of women in the United States who are told that their Papanicolaou (Pap) test was abnormal do not adhere to recommendations for follow-up care. This is a problem especially among minorities and women of lower socioeconomic status. The purpose of this part of the protocol is to test a theory-based intervention designed to improve adherence to follow-up among women who experience an abnormal Pap test. The intervention is a message, delivered over the telephone by a nurse, at the time Pap test results are given to patients. The investigators propose to randomize women who experience an abnormal Pap test to one of three groups: (1) targeted cultural belief + knowledge + importance message (intervention), (2) nontargeted belief + knowledge + importance (active control), or (3) standard care only (passive control). All three groups will receive standard care, which is to notify women by telephone of their abnormal results and provide instructions for follow-up. Women assigned to the intervention group also will receive a cultural belief component consistent with their racial/ethnic group, detailed information about follow-up procedures and the consequences of not returning for follow-up, and information regarding the importance of adhering to recommendations, particularly for "low grade" abnormalities. Women assigned to the active control group will receive a nontargeted belief component, plus procedural knowledge and a message on the importance of follow-up. Adherence to initial follow-up will be the primary outcome. Other behavioral outcomes, such as delayed care and completeness of care, also will be assessed over an 18-month interval by chart review. Additionally, the investigators will evaluate psychological outcomes including anxiety and distress. Finally, the investigators will examine the grade of abnormality (low versus high) as an effect modifier. The investigators anticipate that this research will result in an intervention that will improve several important behavioral and psychological outcomes related to abnormal Pap test results. The intervention is guided by a general integrative theoretical framework; therefore, this research will evaluate an intervention strategy that recognizes the importance of targeting culturally relevant beliefs about follow-up and key determinants of behavior (knowledge/skills, salience, environmental constraints) surrounding abnormal Pap test results. Ultimately, the objective of this research is to improve adherence to follow-up among low-income, minority women who are at particular risk of developing cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 to 55 years who present to the University of Texas Medical Branch (UTMB) clinics for Pap testing.

Exclusion Criteria:

* Women who are currently pregnant
* Have a current diagnosis of cervical cancer; or
* Who are unable to understand English or Spanish.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 341 (Actual)
Dates: Start 2005-10; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carmen R Breitkopf, PhD, Principal Investigator — University of Texas Medical Branch, Galveston
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

REFERENCES:
- [Result] Breitkopf CR, Dawson L, Grady JJ, Breitkopf DM, Nelson-Becker C, Snyder RR. Intervention to improve follow-up for abnormal Papanicolaou tests: a randomized clinical trial. Health Psychol. 2014 Apr;33(4):307-316. doi: 10.1037/a0032722. Epub 2013 Jun 3. PMID 23730719

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Face-to-face recruitment of women 18-55 years of age occurred in 6 University of Texas Medical Branch (UTMB) Regional and Maternal Child Health Program clinics from June 1, 2006-November 30, 2010. Recruitment was interrupted for a period ranging from 2 weeks to 6 months in several clinic sites due to landfall of hurricane Ike on September 13, 2008.
Pre-assignment Details: 6,179 women were eligible during the recruitment period. Of these, 876 declined participation, 4,671 had a normal Pap test result, 254 did not have a Pap test performed at their clinic visit, and 378 had an abnormal Pap test result and could be randomized. Of these, 90% (341/378)were randomized into the 3-arm trial.
Period: Overall Study
Arm/Group | Intervention | Active Control | Standard Care Only
Started | 114 | 114 | 113
Completed | 102 | 101 | 96
Not Completed | 12 | 13 | 17
Not completed — Lost to Follow-up | 4 | 6 | 9
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Clinic Called Patient | 7 | 7 | 7
Not completed — Pregnancy | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Active Control | Standard Care Only | Total
Number analyzed (Participants) | 114 | 114 | 113 | 341
Age, Continuous [Mean (Standard Deviation); unit: years] | 27 (7) | 28 (8) | 29 (8) | 28 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 114 | 114 | 113 | 341
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 114 | 114 | 113 | 341

OUTCOME MEASURES:

1. Primary Outcome: Adherence to Initial Follow-up (Yes/no)
Description: Attendance at initial appointment to follow-up abnormal Pap test result
Time Frame: adherence rates at initial follow-up appointment, 2 weeks to 3 months
Measure: Number; unit: percentage of patients who were adherent
Arm/Group | Intervention | Active Control | Standard Care Only
Number analyzed (Participants) | 102 | 101 | 96
percentage of patients who were adherent | 60 | 54 | 58

2. Secondary Outcome: State Trait Anxiety Inventory (STAI)-State Scale
Description: State Anxiety short form measure (6-item); higher scores =worse outcomes (i.e., higher self-reported anxiety levels)
Time Frame: + 7-30 days post-intervention
Population: Only participants who completed the post-test over the telephone 7-14 following notification of the abnormal Pap test result were asked these questions.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Active Control: non-targeted behavioral and normative beliefs + knowledge/skills + salience + environmental constraints/barriers counseling
  Active control: Partial intervention (full intervention minus cultural-specific component)
Arm/Group | Intervention | Active Control | Standard Care Only
Number analyzed (Participants) | 77 | 76 | 74
units on a scale | 12 (5) | 11 (4) | 11 (4)

ADVERSE EVENTS:
Arm/Group | Intervention | Active Control | Standard Care Only
Serious Adverse Events (participants affected / at risk) | 0/114 | 0/114 | 0/113
Other Adverse Events (participants affected / at risk) | 0/114 | 0/114 | 0/113

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No